CLINICAL TRIAL: NCT03715686
Title: To Accurately Assess Lymph Node Response to Neoadjuvant Chemotherapy by Wire Localization of Clip-marked Axillary Lymph Nodes in Breast Cancer Patients
Brief Title: To Accurately Assess Lymph Node Response to NACT by Wire Localization of Clip-marked Lymph Nodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, director of the department, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BCP24
Record Dates: First submitted 2018-10-13; First posted 2018-10-23 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-09

CONDITIONS: Neoplasm, Breast; Neoadjuvant Chemotherapy; Lymph Node Metastases; Response
Keywords: Neoplasm, Breast; neoadjuvant chemotherapy; Lymph Node Metastases; response
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wire localization (Experimental): Intervention: procedure: wire localization
  Interventions: Procedure: wire localization

INTERVENTIONS:
Procedure: wire localization — Pathologically proven positive axillary lymph node will be clip-marked before the initiation of neoadjuvant chemotherapy. After the completion of neoadjuvant chemotherapy, a wire will be placed to localize the clip-marked node before surgery. During surgery, a standard sentinel lymph node biopsy will be performed as well as the removal of the wire localized node. ALND will be performed in all participants.

SUMMARY:
The investigator developed this protocol to accurately assess lymph node response to neoadjuvant chemotherapy in clinical stage N1 (cN1) breast cancer patients. Accuracy of sentinel lymph node biopsy (SLNB) alone and in combination with the removal of wire-localized-clip-marked nodes will be analyzed. New model to predict lymph node pathological complete remission (pCR) so as to safely avoid axillary lymph node dissection in cN1 breast cancer patients is sought for.

DETAILED DESCRIPTION:
The investigator developed this protocol to accurately assess lymph node response to neoadjuvant chemotherapy in cN1 breast cancer patients. In brief, pathologically proven positive axillary lymph node will be clip-marked before the initiation of neoadjuvant chemotherapy (NACT) and continuously monitored through out the course of chemotherapy with ultrasound. After the completion of neoadjuvant chemotherapy, a wire will be placed to localize the clip-marked node before surgery. During surgery, a standard sentinel lymph node biopsy will be performed as well as the removal of the wire localized node. Axillary lymph node dissection (ALND) will be performed in all participants. Accuracy of SLNB alone and in combination with the removal of wire-localized-clip-marked nodes will be analyzed. Axillary ultrasound and CT scan will be performed before and after neoadjuvant chemotherapy for all patients enrolled. By assessing clinical-pathological and imaging data acquired from this trial, the investigator look forward to developing a model to accurately predict lymph node pCR (AUC >0.85) so as to safely avoid axillary lymph node dissection in cN1 breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* between the age of 18 and 65
* Eastern Cooperative Oncology Group (ECOG) score 0 or 1
* pathologically proven positive axillary lymph node
* enough renal and liver function to sustain chemotherapy
* informed consent obtained

Exclusion Criteria:

* inflammatory breast cancer
* being pregnant or nursing
* neoadjuvant chemotherapy not planned

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of SLNB alone and in combination with the removal of wire-localized-clip-marked nodes. | through study completion, an average of 1 year
  Sensitivity, specificity, false negative rate and negative predictive value will be calculated.

SECONDARY OUTCOMES:
Model to predict lymph node pCR in cN1 patients. | through study completion, an average of 1 year
  Using clinical pathological and image data collected, generate a model to predict lymph node pCR in cN1 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, Dr., Study Director — Beijing Cancer Hosptial
Locations (1):
- Beijing Cancer Hospital Breast Center, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Zheng Q, He Y, Liu Y, Huo L, Zhang N, Wang T, Xie Y, Li J, Ouyang T, Fan Z. Diagnostic accuracy of sentinel lymph node biopsy and wire localized clipped node biopsy after neoadjuvant chemotherapy in node-positive breast cancer. Surg Today. 2025 Feb;55(2):172-179. doi: 10.1007/s00595-024-02981-0. Epub 2024 Dec 27. PMID 39725764